CLINICAL TRIAL: NCT02825225
Title: A Randomized Controlled Trial To Assess and Compare the Outcomes of 20-core Versus 12-core Prostate Biopsy
Brief Title: A Prospective Randomized Trial of Two Different Prostate Biopsy Schemes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Collaborators: Hospital Brigadeiro UGA V-SP (Unknown)
Responsible Party: Principal Investigator, Jose Pontes Jr, MD PhD, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Prostate biopsy - 01
Record Dates: First submitted 2016-06-26; First posted 2016-07-07 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Prostate Cancer; Local Anesthesia; Prostate-Specific Antigen/Blood; Biopsy/Methods; Image-guided Biopsy/Methods; Prostatic Neoplasms/Diagnosis; Prostate/Pathology; Prospective Studies; Humans; Male; Ultrasonography, Interventional/Methods
Keywords: Prostatic Neoplasms; Biopsy; Anesthesia; Detection
MeSH Terms: conditions — Prostatic Neoplasms; Disease | interventions — Alkalies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 20 core-biopsy fragments (Experimental): Patients submitted to experimental intervention (extended sextant biopsy with 20 cores) compared to current standard biopsy protocol (extended sextant biopsy with 12 cores) guided by transrectal ultrasound.
  Interventions: Other: 20 core-biopsy fragments; Procedure: Base and apex local anesthesia
- Base and apex local anesthesia (Experimental): Patients submitted to experimental intervention in prostate-biopsy anesthetic protocol (prostate base and prostate apex bilateral local anesthetic injection) compared to participants submitted to current standard anesthetic protocol in institution (prostate base bilateral local anesthesia) guided by transrectal ultrasound. guided by transrectal ultrasound.
  Interventions: Other: 20 core-biopsy fragments; Procedure: Base and apex local anesthesia

INTERVENTIONS:
Other: 20 core-biopsy fragments — Using the extended sextant fashion prostate biopsy, this randomized group was submitted to a 20-fragments core-biopsy to evaluate the diagnostic power, pain perception and complications comparative to institution's standard 12 cores.
Procedure: Base and apex local anesthesia — Using the institution's standard local anesthesia protocol (base injection) as active comparator group, this randomized group was submitted to base and apex local anesthetic application to evaluate tolerability of the procedure, pain perception (with use of previous validated analogue pain scale) and complications.

SUMMARY:
The main purpose is to compare the detection rate of 20-core versus 12-core prostate biopsy. The secondary objective is to evaluate pain perception using a validated scale to compare the analgesia provided by the two different local anesthesia schemes. Data will be prospectively collected from patients who will undergo prostate biopsy in a single high volume urology center. The patients will be randomized to two different biopsy samplings and two local anesthesia schemes.

DETAILED DESCRIPTION:
Prostate cancer is male's leading solid non-cutaneous tumor, and the second cause of cancer death in western countries. The main risk factors are age (5th decade or more), family history and life-style (low physical activity and occidental dietary habit). Due to it's high incidence and mortality, the screening protocols continue to be supported worldwide by the urologic and oncologic societies. The diagnosis of this disease needs histological evidence that is obtained by prostate biopsy which is indicated when prostate specific antigen (PSA) serum levels are elevated or there is suspicion at digital rectal examination. Actual estimations conclude that more than 200.000 new cases are diagnosed per-year in US and much more patients are submitted to biopsies; turning prostate biopsy a routine medical procedure. In therms of current medical evidence there is controversy in some biopsy aspects. The ideal number of fragments to be obtained is not well established. While twelve core is believed to be the minimum to be sampled, the maximum number is not clear. To ease the estimation of the number of necessary core at biopsy the literature recommend the use of nomograms; they adequate the number of removed fragments according to each individual characteristics such as age, volume, previous biopsy and PSA levels. The prostate biopsy is considered a painful procedure by 96% of patients, therefore it is fundamental to soften the soreness employing some form of anesthesia. There is no consensus regarding the ideal protocol but the local anesthesia with the periprostatic blockade is the most employed worldwide. However there is a controversy related to the site of the injection during the periprostatic block in terms of efficacy: base versus apex or both sites.

Considering the epidemiological importance of prostate cancer detection in a continuous aging population, this study protocol was enrolled in a single center high volume urology Brazilian Public Hospital. The patients will be randomized at a 1:1 ratio for the two biopsy schemes and for the two anesthesia templates.The main objective was to compare the detection rate of two different prostate biopsy schemes 20-core versus 12-core prostate biopsy guided by transrectal ultrasound. Secondary objectives were to evaluate pain perception of the two local anesthesia schemes using a validated pain scale. The pain was evaluated using the visual pain scale immediately after the biopsy and one hour after the procedure. The patients were contacted by phone one week after the biopsy to assess the occurrence of any complication. The investigators then compared the major and minor complication rates of 20-core versus 12-core protocol using the Clavien-Dindo scale. In those patients with cancer at the pathologic report that underwent radical prostatectomy, the investigators will also compare the concordance of Gleason score between the biopsy versus surgical specimen according to the biopsy scheme 20-core versus 12-core.

Data was collected since mid 2012 up to june 2016, inclusion and exclusion criteria will be detailed elsewhere. All information was obtained by the main investigator and all procedures were supervised by the main investigator as well.

ELIGIBILITY:
Inclusion Criteria:

* Formal indication to prostate biopsy: PSA elevation, positive digital rectal examination of prostate, prostate cancer active surveillance protocols.
* Patients signing the consent therm agreeing to participate in the trial
* Exclusive local anesthesia prostate biopsy.
* Exclusive transrectal ultrasound guided prostate biopsy.

Exclusion Criteria:

* Transperineal ultrasound guided prostate biopsy
* Magnetic resonance cognitive fusion biopsy.
* Previous treatment with radiation therapy or brachytherapy.
* Previous treatment with focal therapy
* Previous androgen deprivation therapy

Min Age: 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Actual)
Dates: Start 2012-05; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with prostate cancer detected. | Through study completion, an average of four years.
  Statistical evaluation comparing detection of prostate cancer in 12-core versus 20 cores.

SECONDARY OUTCOMES:
Number of participants with complications | Immediate, early (30 minutes) and late (within first week)
  Comparison of data between 12 versus 20 core-biopsy and base versus base plus apex anesthesia in therms of complication occurrence.
Core biopsy accuracy. | Through study completion, at time of surgery.
  Comparison of cancer positive pathology data between 12 and 20 core-biopsy with their respective radical prostatectomy hole mount pathology specimen (when treatment was indicated).
Pain perception using pain analogue scale. | Immediate and early (30 minutes after biopsy).
  Compare pain perception of two anesthesia scheme base versus base plus apex using the visual pain analogue scale immediately after the biopsy and 30 minutes later. The investigators will also compared the analgesia of these schemes according to PSA, PSA density, free/total PSA ratio, prostate volume, previous biopsy.
Number of participants with prostate cancer detected according to PSA value | Through study completion, an average of four years.
  The investigators will also compare the detection rate of 12 versus 20 fragments schemes according to the PSA value.
Number of participants with prostate cancer detected according to PSA density. | Through study completion, an average of four years.
  The investigators will also compare the detection rate of 12 versus 20 fragments schemes according to the PSA density.
Number of participants with prostate cancer detected according to free/total PSA ratio. | Through study completion, an average of four years.
  The investigators will also compare the detection rate of 12 versus 20 fragments schemes according to the PSA free/total PSA ratio.
Number of participants with prostate cancer detected according to prostate volume. | Through study completion, an average of four years.
  The investigators will also compare the detection rate of 12 versus 20 fragments schemes according to prostate volume.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Pontes Jr, MD PhD, Principal Investigator — University of Nove de Julho
Locations (1):
- Hospital Brigadeiro UGA V-SP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
Secrecy will be maintained in observation of ethics committee opinion.

REFERENCES:
- [Result] Siegel R, DeSantis C, Virgo K, Stein K, Mariotto A, Smith T, Cooper D, Gansler T, Lerro C, Fedewa S, Lin C, Leach C, Cannady RS, Cho H, Scoppa S, Hachey M, Kirch R, Jemal A, Ward E. Cancer treatment and survivorship statistics, 2012. CA Cancer J Clin. 2012 Jul-Aug;62(4):220-41. doi: 10.3322/caac.21149. Epub 2012 Jun 14. PMID 22700443
- [Result] Giovannucci E, Liu Y, Platz EA, Stampfer MJ, Willett WC. Risk factors for prostate cancer incidence and progression in the health professionals follow-up study. Int J Cancer. 2007 Oct 1;121(7):1571-8. doi: 10.1002/ijc.22788. PMID 17450530
- [Result] Crawford ED. Epidemiology of prostate cancer. Urology. 2003 Dec 22;62(6 Suppl 1):3-12. doi: 10.1016/j.urology.2003.10.013. PMID 14706503
- [Result] Schroder FH, Hugosson J, Roobol MJ, Tammela TL, Ciatto S, Nelen V, Kwiatkowski M, Lujan M, Lilja H, Zappa M, Denis LJ, Recker F, Paez A, Maattanen L, Bangma CH, Aus G, Carlsson S, Villers A, Rebillard X, van der Kwast T, Kujala PM, Blijenberg BG, Stenman UH, Huber A, Taari K, Hakama M, Moss SM, de Koning HJ, Auvinen A; ERSPC Investigators. Prostate-cancer mortality at 11 years of follow-up. N Engl J Med. 2012 Mar 15;366(11):981-90. doi: 10.1056/NEJMoa1113135. PMID 22417251
- [Result] Ross AE, Loeb S, Landis P, Partin AW, Epstein JI, Kettermann A, Feng Z, Carter HB, Walsh PC. Prostate-specific antigen kinetics during follow-up are an unreliable trigger for intervention in a prostate cancer surveillance program. J Clin Oncol. 2010 Jun 10;28(17):2810-6. doi: 10.1200/JCO.2009.25.7311. Epub 2010 May 3. PMID 20439642
- [Result] Thompson IM, Goodman PJ, Tangen CM, Lucia MS, Miller GJ, Ford LG, Lieber MM, Cespedes RD, Atkins JN, Lippman SM, Carlin SM, Ryan A, Szczepanek CM, Crowley JJ, Coltman CA Jr. The influence of finasteride on the development of prostate cancer. N Engl J Med. 2003 Jul 17;349(3):215-24. doi: 10.1056/NEJMoa030660. Epub 2003 Jun 24. PMID 12824459
- [Result] Zisman A, Leibovici D, Kleinmann J, Siegel YI, Lindner A. The impact of prostate biopsy on patient well-being: a prospective study of pain, anxiety and erectile dysfunction. J Urol. 2001 Feb;165(2):445-54. doi: 10.1097/00005392-200102000-00023. PMID 11176394
- [Result] Nash PA, Bruce JE, Indudhara R, Shinohara K. Transrectal ultrasound guided prostatic nerve blockade eases systematic needle biopsy of the prostate. J Urol. 1996 Feb;155(2):607-9. PMID 8558671
- [Result] Rodriguez-Covarrubias F, Gonzalez-Ramirez A, Aguilar-Davidov B, Castillejos-Molina R, Sotomayor M, Feria-Bernal G. Extended sampling at first biopsy improves cancer detection rate: results of a prospective, randomized trial comparing 12 versus 18-core prostate biopsy. J Urol. 2011 Jun;185(6):2132-6. doi: 10.1016/j.juro.2011.02.010. Epub 2011 Apr 15. PMID 21496851
- [Result] Sfakianos JP, Thorner DA, Dovirak O, Weiss JP, Karanikolas NT. Optimizing prostate cancer detection during biopsy by standardizing the amount of tissue examined per core. BJU Int. 2011 Nov;108(10):1578-81. doi: 10.1111/j.1464-410X.2011.10239.x. Epub 2011 May 31. PMID 21627750
- [Result] Remzi M, Fong YK, Dobrovits M, Anagnostou T, Seitz C, Waldert M, Harik M, Marihart S, Marberger M, Djavan B. The Vienna nomogram: validation of a novel biopsy strategy defining the optimal number of cores based on patient age and total prostate volume. J Urol. 2005 Oct;174(4 Pt 1):1256-60; discussion 1260-1; author reply 1261. doi: 10.1097/01.ju.0000173924.83392.cc. PMID 16145388
- [Result] Zaytoun OM, Jones JS. Prostate cancer detection after a negative prostate biopsy: lessons learnt in the Cleveland Clinic experience. Int J Urol. 2011 Aug;18(8):557-68. doi: 10.1111/j.1442-2042.2011.02798.x. Epub 2011 Jun 21. PMID 21692866
- [Result] Ukimura O, Coleman JA, de la Taille A, Emberton M, Epstein JI, Freedland SJ, Giannarini G, Kibel AS, Montironi R, Ploussard G, Roobol MJ, Scattoni V, Jones JS. Contemporary role of systematic prostate biopsies: indications, techniques, and implications for patient care. Eur Urol. 2013 Feb;63(2):214-30. doi: 10.1016/j.eururo.2012.09.033. Epub 2012 Sep 25. PMID 23021971
- [Result] Pepe P, Aragona F. Saturation prostate needle biopsy and prostate cancer detection at initial and repeat evaluation. Urology. 2007 Dec;70(6):1131-5. doi: 10.1016/j.urology.2007.07.068. PMID 18158033
- [Result] Sonn GA, Natarajan S, Margolis DJ, MacAiran M, Lieu P, Huang J, Dorey FJ, Marks LS. Targeted biopsy in the detection of prostate cancer using an office based magnetic resonance ultrasound fusion device. J Urol. 2013 Jan;189(1):86-91. doi: 10.1016/j.juro.2012.08.095. Epub 2012 Nov 14. PMID 23158413
- [Result] King CR, McNeal JE, Gill H, Presti JC Jr. Extended prostate biopsy scheme improves reliability of Gleason grading: implications for radiotherapy patients. Int J Radiat Oncol Biol Phys. 2004 Jun 1;59(2):386-91. doi: 10.1016/j.ijrobp.2003.10.014. PMID 15145152
- [Result] Descazeaud A, Rubin M, Chemama S, Larre S, Salomon L, Allory Y, Vordos D, Hoznek A, Yiou R, Chopin D, Abbou C, de la Taille A. Saturation biopsy protocol enhances prediction of pT3 and surgical margin status on prostatectomy specimen. World J Urol. 2006 Dec;24(6):676-80. doi: 10.1007/s00345-006-0134-7. Epub 2006 Nov 7. PMID 17089179
- [Result] Marks LS, Fradet Y, Deras IL, Blase A, Mathis J, Aubin SM, Cancio AT, Desaulniers M, Ellis WJ, Rittenhouse H, Groskopf J. PCA3 molecular urine assay for prostate cancer in men undergoing repeat biopsy. Urology. 2007 Mar;69(3):532-5. doi: 10.1016/j.urology.2006.12.014. PMID 17382159
- [Result] Leite KR, Tomiyama A, Reis ST, Sousa-Canavez JM, Sanudo A, Dall'Oglio MF, Camara-Lopes LH, Srougi M. MicroRNA-100 expression is independently related to biochemical recurrence of prostate cancer. J Urol. 2011 Mar;185(3):1118-22. doi: 10.1016/j.juro.2010.10.035. Epub 2011 Jan 21. PMID 21255804
- [Result] Leite KR, Sousa-Canavez JM, Reis ST, Tomiyama AH, Camara-Lopes LH, Sanudo A, Antunes AA, Srougi M. Change in expression of miR-let7c, miR-100, and miR-218 from high grade localized prostate cancer to metastasis. Urol Oncol. 2011 May-Jun;29(3):265-9. doi: 10.1016/j.urolonc.2009.02.002. Epub 2009 Apr 16. PMID 19372056
- See also: European society of Urology guidelines on prostate cancer — http://www.uroweb.org/guidelines/online-guidelines/